CLINICAL TRIAL: NCT07377825
Title: Accuracy and Periodontal Outcomes of Three Interproximal Enamel Reduction Techniques During Clear Aligner Therapy: A Randomized Controlled Trial
Brief Title: Accuracy and Periodontal Outcomes of Three Interproximal Enamel Reduction Techniques During Clear Aligner Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Omar Alkadhi, Associate Professor of Orthodontics, Riyadh Elm University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REU-IPR-CAT-RCT-2026-001
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Dental Crowding,Interproximal Enamel Reduction; Malocclusion, Angle's Class; Periodontal Diseases
Keywords: Clear Aligner Therapy; Periodontal Disease; Interproximal Enamel Reduction
MeSH Terms: conditions — Crowding; Malocclusion; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Three-arm, parallel-group, superiority randomized controlled trial. Participants undergoing clear aligner therapy with IPR prescribed will be randomized 1:1:1 to manual arm, motor-driven arm, or abrasive arm. IPR accuracy will be assessed using intraoral scans before and immediately after IPR; periodontal indices will be assessed at baseline and 6-week follow-up
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual arm (Experimental): Interproximal enamel reduction will be performed at the prescribed contacts using manual abrasive strips (6 mm separating abrasive strips, coarse; Ortho Organizers, Inc., Carlsbad, USA). (n = 25)
  Interventions: Procedure: Manual Arm
- Motor-driven arm (Experimental): Interproximal enamel reduction will be performed at the prescribed contacts using motor-driven oscillating strips (OK Strips Kit with JAINTEK EVA handpiece operated at < 15,000 rpm; JAINTEK Co., Ltd., Guri-si, Republic of Korea). (n = 25).
  Interventions: Procedure: Motor Driven Arm
- Abrasive arm (Experimental): Interproximal enamel reduction will be performed at the prescribed contacts using abrasive discs (OK DIA DISC, double-sided, thickness 0.15 mm; JAINTEK Co., Ltd., Guri-si, Republic of Korea). (n = 25).
  Interventions: Procedure: Abrasive Arm

INTERVENTIONS:
Procedure: Manual Arm — Interproximal enamel reduction (IPR) will be performed at the contacts prescribed in the participant's digital treatment plan using manual abrasive strips (6 mm separating abrasive strips, coarse; Ortho Organizers, Inc., Carlsbad, USA). IPR will be performed by the same trained and calibrated operator, and interproximal clearance will be verified using metal interproximal gauges
  Arms: Manual arm
Procedure: Motor Driven Arm — Interproximal enamel reduction will be performed at the prescribed contacts using motor-driven oscillating strips (OK Strips Kit with JAINTEK EVA handpiece operated at < 15,000 rpm; JAINTEK Co., Ltd., Guri-si, Republic of Korea). IPR will be performed by the same trained and calibrated operator and interproximal clearance will be verified using metal interproximal gauges. (n = 25)
  Arms: Motor-driven arm
Procedure: Abrasive Arm — Interproximal enamel reduction will be performed at the prescribed contacts using abrasive discs (OK DIA DISC, double-sided, thickness 0.15 mm; JAINTEK Co., Ltd., Guri-si, Republic of Korea). IPR will be performed by the same trained and calibrated operator and interproximal clearance will be verified using metal interproximal gauges. (n = 25)
  Arms: Abrasive arm

SUMMARY:
This randomized controlled clinical trial will compare three commonly used interproximal enamel reduction (IPR) techniques during clear aligner therapy in adult patients. IPR is a routine orthodontic procedure in which a small amount of enamel is removed between teeth to create space and help achieve the planned alignment.

Seventy-five adults (18 years and older) indicated for receiving clear aligner treatment with IPR prescribed in their digital treatment plan will be enrolled at the orthodontic clinics of Riyadh Elm University (Riyadh, Saudi Arabia) and randomized in a 1:1:1 ratio to one of three IPR techniques: manual abrasive strips (manual arm), motor-driven oscillating strips (motor-driven arm), or abrasive discs (abrasive arm). IPR will be performed by the same trained operator according to the assigned technique.

The primary outcome is IPR accuracy, defined as the difference between the amount of IPR planned digitally and the amount performed clinically, measured using intraoral scans taken before and immediately after IPR. Secondary outcomes are short-term periodontal outcomes, assessed on IPR teeth only using plaque and gingival bleeding indices at baseline and at a 6-week follow-up visit. The data analyst will be blinded to group allocation

DETAILED DESCRIPTION:
2.1. Aim This study aims to compare, in patients undergoing clear aligner therapy, the accuracy of interproximal enamel reduction (IPR) and the short term periodontal effects among three techniques: manual hand strips, motor driven oscillating strips, and abrasive discs.

2.2 Objectives

1. To Quantify and compare the accuracy of interproximal enamel reduction among manual hand strips, motor driven oscillating strips, and abrasive discs during clear aligner therapy.
2. To Evaluate and compare the short term periodontal effects of IPR among manual hand strips, motor driven oscillating strips, and abrasive discs
3. Hypothesis and/ or Research Question:

   There is no difference between manual hand strips, motor driven oscillating strips, and abrasive discs in the accuracy of interproximal enamel reduction and in the short term changes in plaque index and bleeding on probing.
4. Materials and Methods:

   4.1. Study Design This study will be a single-blinded randomized controlled clinical trial with three parallel arms and equal allocation of 1:1:1 conducted at the orthodontic clinics of Riyadh Elm University, Riyadh, Saudi Arabia. The trial will be registered at ClinicalTrials.gov and approval will be obtained from the Saudi Food and Drug Authority with ethical approval from Riyadh Elm University Institutional Review Board (IRB).

   4.2. Sample size Sample size calculation was performed using GPower (version 3.1.9.6). Based on data reported by Hariharan et al. (2022), a large effect size (Cohen's f = 0.40) was assumed for differences in the accuracy of interproximal reduction between three techniques. With a significance level of 0.05 and a power of 80%, a total sample size of 66 patients was required. Allowing for a 10% dropout rate, 75 patients (25 per group) were planned.

   4.3. Study Participants and Experiment:

   a. Participants: Adult patients receiving Lite, Moderate or Comprehensive Invisalign® treatment packages (Align Technology, Inc., San Jose, CA, USA) at the orthodontic clinics of Riyadh Elm University, Riyadh, Saudi Arabia, will be screened at the pre treatment visit or at the first scheduled IPR appointment. Eligible patients who provide written informed consent will be enrolled in this study.

   Eligibility Criteria

   Inclusion criteria Exclusion criteria Age 18 years or older with full permanent dentition orthodontic treatment plan including extraction

   Undergoing clear aligner therapy with Invisalign® with a ClinCheck™ treatment plan that includes interproximal enamel reduction Proximal restorations or caries on any tooth surface targeted for interproximal enamel reduction.

   Periodontally healthy patient Current smoking, diabetes mellitus, or other systemic diseases known to affect periodontal status

   Exclusion criteria orthodontic treatment plan including extraction

   Proximal restorations or caries on any tooth surface targeted for interproximal enamel reduction.

   Current smoking, diabetes mellitus, or other systemic diseases known to affect periodontal status

   4.4. Randomization and allocation concealment: Group assignment will use simple randomization in a 1:1:1 ratio generated via a secure web-based random sequence tool. An independent coordinator will prepare a master Excel list linking unique serial numbers (e.g., 001, 002, …) to the three trial arms according to that sequence. Each number will be printed on an identical, opaque ticket. At enrolment, a trained dental assistant will present an opaque draw bowl containing the prepared tickets; the participant will draw one number. The dental assistant will record the patient ID and drawn number in the allocation log and contact the independent coordinator to obtain the corresponding assignment. Used tickets will be retained and not returned to the bowl.

   4.5. Intervention: At the IPR visit, an intraoral scan will be acquired using the iTero Element 5D (Align Technology, Inc., San Jose, CA, USA) dental plaque will be assessed using the Plaque Index of Silness and Löe (1964) on teeth scheduled to receive IPR only. Baseline periodontal assessment will be performed only on the teeth scheduled to receive IPR, including Plaque Index (Silness & Löe, 1964), and Gingival Bleeding Index (Ainamo & Bay, 1975).

   IPR will then be performed at the contacts as prescribed in the ClinCheck treatment plan by the same trained and calibrated operator according to the allocated technique. Interproximal clearance will be verified using metal interproximal gauges. A second intraoral scan will be acquired immediately after IPR during the same visit (T1). At 6 weeks after IPR, participants will be recalled and periodontal reassessment will be performed on the same IPR teeth only, using: Plaque Index (Silness & Löe, 1964), and Gingival Bleeding Index (Ainamo & Bay, 1975). No polishing and no topical fluoride will be used in any study group.

   Group 1 Manual abrasive strips will be used, specifically 6 mm Separating Abrasive Strips (coarse) (Ortho Organizers, Inc.).

   Group 2 Motor driven oscillating strips will be used, specifically the OK Strips KIT with a JAINTEK EVA Ahandpiece operated at less than 15,000 rpm.

   Group 3 Oscillating segmented discs will be used, specifically Komet oscillating segmented OS discs (OS1Mm).

   4.6. Outcomes and measurements

   Standard Tessellation Language (STL) files will be exported from the iTero platform and imported into OrthoCAD digital software version 5.9.0.36 (3Shape, Copenhagen, Denmark), which will be used to measure the widest mesiodistal diameter of each incisor, canine, and premolar scheduled to receive IPR at baseline before IPR (T0) and immediately after IPR (T1); the amount of IPR performed will be calculated as the difference in the summed mesiodistal widths of the IPR teeth between T0 and T1 and will be compared with the planned IPR values extracted from the initial ClinCheck treatment plan. Periodontal parameters will be assessed on IPR teeth only and compared between baseline and the 6-week follow-up: bleeding on probing will be assessed at six sites per tooth using gentle probing force of approximately 25 g and scored as 0 for absence of bleeding and 1 for presence of bleeding within 10-15 seconds, and plaque will be assessed using the Plaque Index of Silness and Löe (1964) on four surfaces per tooth with scores summed and divided by four to obtain the tooth-level plaque index To assess intra examiner reliability of the OrthoCAD mesiodistal width measurements, a random subsample of 20 participants will be re measured by the same operator after a 2 week interval under identical conditions.
5. Statistical analysis Statistical analysis will be performed using SPSS software (Version 26.0; IBM Corp, Armonk, NY). Descriptive statistics, including means and standard deviations for normally distributed data, or medians and interquartile ranges for non-parametric data, will be calculated for all variables.

   Intra-examiner reliability for mesiodistal width measurements will be assessed using the Intraclass Correlation Coefficient (ICC) with 95% confidence intervals based on the remeasurement of 20 randomly selected participants.

   The Shapiro-Wilk test will be used to assess the normality of the data. For the primary outcome (IPR accuracy), if a normal distribution is confirmed, a One-Way Analysis of Variance (ANOVA) will be used to compare the three groups, followed by Tukey's HSD post-hoc test for pairwise comparisons. If normality is violated, the Kruskal-Wallis test with Bonferroni adjustment will be employed.

   For periodontal measurements (Plaque Index and Gingival Bleeding Index), changes between baseline (T0) and 6-week follow-up (T1) within each group will be analyzed using the Wilcoxon signed-rank test. Comparisons of these changes among the three intervention groups will be conducted using the Kruskal-Wallis test. The level of significance for all tests will be set at p<0.05.
6. Ethical considerations:

Ethical approval will be obtained from Riyadh Elm University Institutional Review Board (IRB) and approval will be obtained from the Saudi Food and Drug Authority as applicable. The trial will be registered on ClinicalTrials.gov before recruitment. Written informed consent will be obtained from all participants. Participants may withdraw at any time without affecting their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older with full permanent dentition.
* Undergoing clear aligner therapy (Invisalign) with a ClinCheck treatment plan that includes interproximal enamel reduction (IPR).
* Periodontally healthy at baseline (per clinic screening).

Exclusion Criteria:

* Orthodontic treatment plan including extractions.
* Proximal restorations or caries on any tooth surface targeted for IPR.
* Current smoking.
* Diabetes mellitus or other systemic diseases known to affect periodontal status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Accuracy of interproximal enamel reduction (IPR) (planned vs performed, mm) | Baseline (pre-IPR intraoral scan) to immediately after IPR (post-IPR intraoral scan), same visit
  Planned IPR (mm) will be extracted from the participant's initial digital treatment plan (ClinCheck) for the contacts scheduled for IPR at the study visit. Performed IPR (mm) will be quantified using intraoral scans obtained immediately before and immediately after IPR. STL files will be analyzed in OrthoCAD to measure the mesiodistal tooth widths of incisors, canines, and premolars receiving IPR. The amount of performed IPR will be calculated as the difference in the summed mesiodistal widths of the included teeth before vs after IPR (pre-IPR minus post-IPR). IPR accuracy will be calculated per participant as the discrepancy between planned and performed IPR (mm) and compared across the three groups.

SECONDARY OUTCOMES:
Changes in plaque Index | Baseline (pre-IPR) to 6 weeks after IPR.
  Plaque will be assessed using the Plaque Index of Silness and Löe (1964) on four surfaces per tooth with scores summed and divided by four to obtain the tooth-level plaque index
Changes in gingival bleeding index | Baseline (pre-IPR) to 6 weeks after IPR.
  Bleeding on probing will be assessed at six sites per tooth using gentle probing force of approximately 25 g and scored as 0 for absence of bleeding and 1 for presence of bleeding within 10-15 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: omar alkadhi, Principal Investigator — Riyadh Elm University; Abdulwahab Ahmed Alamri, Principal Investigator — Riyadh Elm University
Locations (1):
- Riyadh Elm University, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shalchi M, Abdollahi N, Shafiei Haghshenas E, Khabbaz S, Olyaee P. Effect of Interdental Enamel Reduction on Clinical Attachment Loss, Bleeding on Probing, and Incidence of Caries in Treating Class I Malocclusion Cases: A Retrospective Cohort Study. Cureus. 2023 Feb 15;15(2):e35018. doi: 10.7759/cureus.35018. eCollection 2023 Feb. PMID 36938231
- [Background] Gulec Ergun P, Arman Ozcirpici A, Atakan Kocabalkan A, Tuncer NI. Evaluation of the Consistency of Two Interproximal Reduction Methods in Clear Aligner Therapy: A Preliminary Study. Turk J Orthod. 2024 Mar 28;37(1):1-6. doi: 10.4274/TurkJOrthod.2023.2022.158. PMID 38556946
- [Background] Gulec-Ergun P, Arman-Ozcirpici A, Atakan-Kocabalkan A, Tuncer NI. Comparison of the accuracy of three interproximal reduction methods used in clear aligner treatment. Clin Oral Investig. 2024 Jan 15;28(1):95. doi: 10.1007/s00784-024-05499-4. PMID 38221544
- [Background] Kalemaj Z, Levrini L. Quantitative evaluation of implemented interproximal enamel reduction during aligner therapy. Angle Orthod. 2021 Jan 1;91(1):61-66. doi: 10.2319/040920-272.1. PMID 33339043
- [Background] Fiori A, Minervini G, Nucci L, d'Apuzzo F, Perillo L, Grassia V. Predictability of crowding resolution in clear aligner treatment. Prog Orthod. 2022 Nov 28;23(1):43. doi: 10.1186/s40510-022-00438-z. PMID 36437397
- [Background] Lagana G, Malara A, Lione R, Danesi C, Meuli S, Cozza P. Enamel interproximal reduction during treatment with clear aligners: digital planning versus OrthoCAD analysis. BMC Oral Health. 2021 Apr 19;21(1):199. doi: 10.1186/s12903-021-01487-2. PMID 33874922
- [Background] Hariharan A, Arqub SA, Gandhi V, Da Cunha Godoy L, Kuo CL, Uribe F. Evaluation of interproximal reduction in individual teeth, and full arch assessment in clear aligner therapy: digital planning versus 3D model analysis after reduction. Prog Orthod. 2022 Mar 7;23(1):9. doi: 10.1186/s40510-022-00403-w. PMID 35254555
- [Background] De Felice ME, Nucci L, Fiori A, Flores-Mir C, Perillo L, Grassia V. Accuracy of interproximal enamel reduction during clear aligner treatment. Prog Orthod. 2020 Jul 28;21(1):28. doi: 10.1186/s40510-020-00329-1. PMID 32719906